CLINICAL TRIAL: NCT05759637
Title: Type 2 Diabetes, Obesity and Cortisol Excess
Acronym: DOCOR
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Siena (Other); Niguarda Hospital (Other); Campus Bio-Medico University (Other); Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Italy (Other)
Responsible Party: Sponsor
Other Study IDs: 05J101
Record Dates: First submitted 2023-02-26; First posted 2023-03-08 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Cortisol; Hypersecretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- T2D: patients with Type2 diabetes (T2D)
  Interventions: Diagnostic Test: 1mg DST
- obese without T2D: obese patients without Type 2 diabetes (T2D)
  Interventions: Diagnostic Test: 1mg DST

INTERVENTIONS:
Diagnostic Test: 1mg DST — measurement of cortisol levels after 1 mg of dexamethasone (DST) at 11 pm

SUMMARY:
The present observational cross-sectional study is aimed to assess: the hidden hypercortisolism (HidHyCo) prevalence in a sample of Type 2 diabetes (T2D) patients and the clinical characteristics more frequently associated with the HidHyCo presence and the HidHyCo prevalence in an adequate sample of obese patients without T2D and the clinical characteristics more frequently associated with the HidHyCo presence.

DETAILED DESCRIPTION:
Mild and asymptomatic hypercortisolism has been described to be associated with increased prevalence of chronic complications of cortisol excess, such as osteoporosis, hypertension, type 2 diabetes (T2D) and obesity and with increased mortality. In patients with osteoporosis, hypertension, T2D or obesity, this form of hypercortisolism may remain occult (hidden hypercortisolism, HidHyCo), until its presence is suspected on the basis of particular characteristics of the underlying diseases. The HidHyCo prevalence in the general population is estimated to be 0.2-2%, but it has been suggested to be even higher (up to 10%) in some specific populations as for example in patients T2D. Data regarding the prevalence of HidHyCo in obese populations are limited, Therefore, the issue of which diabetic or obese patient has to be screened for HidHyCo has recently become a widely debated topic. Therefore, the aims of the present study protocol are to assess: i) the HidHyCo prevalence in a sample of T2D patients and the clinical characteristics more frequently associated with the HidHyCo presence; ii) the HidHyCo prevalence in an adequate sample of obese patients without T2D and the clinical characteristics more frequently associated with the HidHyCo presence.

All T2D and obese-without T2D patients between 18 and 75 years of age, consecutively referred to the out-patient clinics for Diabetes and Obesity of our center will be assessed for possible inclusion. At the enrolment in all patients anthropometric e biochemical variables will be recorded. At the enrolment we will evaluate cortisol levels after dexamethasone suppression test (F-1mgDST) in all T2D and obese-without T2D patients, who have been included in the study and who have given the informed consent to participate in the study. In all subjects with F-1mgDST >1.8 μg/dL, cortisol levels after two-day low dose (2 mg/day) dexamethasone suppression test (F-2mgx2dDST) will be performed. Patients with F-2mgx2dDST above >1.8 μg/dL will be considered affected with possible HidHyCo and will be studied following the available guidelines for the diagnosis of hypercortisolism.

ELIGIBILITY:
Inclusion Criteria:

patients with T2D and Obesity

Exclusion Criteria:

* pregnancy/breast feeding,
* sleep apnea,
* prepuberal onset of hypertension, hormonal hypersecreting adrenal mass,
* symptoms of hypercortisolism;
* already known secondary hypertension;
* conditions associated with increased hypothalamic-pituitary-adrenal (HPA) axis activity, -severe autoimmune/rheumatologic and hematologic diseases, alcoholism, kidney disease (glomerular filtration rate <60)
* drugs influencing the HPA axis activity. For inclusion in Group 2 the presence of T2D will be an exclusion criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All T2D and obese patients between 18 and 75 years of age, consecutively referred to the out-patient clinics for Diabetes and Obesity of our center
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2025-12-06 (Estimated); Study Completion 2025-12-06 (Estimated)

PRIMARY OUTCOMES:
Hidden Hypercortisolism prevalence in a sample of T2D patients | 24 months
  prevalence of patients with F-1mgDST>1.8 mcg/dl
Hidden Hypercortisolism prevalence in a sample of Obese patients | 24 months
  prevalence of patients with F-1mgDST>1.8 mcg/dl

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Istituto Auxologico Italiano, Milan
  - Niguarda Hospital, Milan
  - Campus Bio-Medico University, Roma
  - University of Siena, Siena
  - Azienda Ospedaliero Universitaria, Santa Maria della Misericordia di Udine, Udine